CLINICAL TRIAL: NCT01926782
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of an Every Four Weeks Treatment Regimen of Alirocumab in Patients With Primary Hypercholesterolemia
Brief Title: Study to Evaluate the Efficacy and Safety of an Every Four Weeks Treatment Regimen of Alirocumab (REGN727/ SAR236553) in Patients With Primary Hypercholesterolemia (ODYSSEY CHOICE 1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R727-CL-1308
Record Dates: First submitted 2013-08-19; First posted 2013-08-21 (Estimated); Results first posted 2017-03-21 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-01

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — alirocumab; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Intervention Model Description: The study was conducted in 2 separate populations concurrently: subjects receiving concomitant statin therapy and subjects not receiving concomitant statin therapy. Subjects receiving concomitant statin were to receive stable daily doses of rosuvastatin, atorvastatin, or simvastatin for at least 4 weeks. Background treatment with other lipid-modifying therapy (LMT) was allowed for all patients, provided they had been on a stable dose for at least 4 weeks (6 weeks for fenofibrate) prior to study entry.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo Q2W (Placebo Comparator): Two subcutaneous (SC) injections of placebo (for alirocumab) Q2W with or without stable statin therapy for 48 weeks.
  Interventions: Drug: Placebo (for alirocumab); Drug: Statin
- Alirocumab 75 mg/ Up 150 mg Q2W (Experimental): One SC injection of each Alirocumab 75 mg and placebo Q2W with or without stable statin therapy for 48 weeks. Alirocumab dose up-titrated to 150 mg from Week 12 when LDL-C levels ≥ 70 mg/dL (1.81 mmol/L) (for very high CV risk participants) or ≥ 100 mg/dL (2.59 mmol/L) (for moderate and high CV risk participants) at Week 8.
  Interventions: Drug: Placebo (for alirocumab); Drug: Alirocumab; Drug: Statin
- Alirocumab 300 mg/ Up 150 mg Q4W (Experimental): Two SC injections of Alirocumab 150 mg Q4W alternating with two SC injections of placebo Q4W with or without stable statin therapy for 48 weeks. Alirocumab dose up-titrated to 150 mg from Week 12 when LDL-C levels ≥ 70 mg/dL (1.81 mmol/L) (for very high CV risk participants) or ≥ 100 mg/dL (2.59 mmol/L) (for moderate and high CV risk participants) at Week 8.
  Interventions: Drug: Placebo (for alirocumab); Drug: Alirocumab; Drug: Statin

INTERVENTIONS:
Drug: Placebo (for alirocumab) — Solution for injection, subcutaneous injections in the abdomen, thigh, or outer area of upper arm with an auto-injector.
Drug: Alirocumab — Solution for injection, subcutaneous injection in the abdomen, thigh, or outer area of upper arm with an auto-injector.
  Other Names: SAR236553; REGN727; Praluent
  Arms: Alirocumab 300 mg/ Up 150 mg Q4W; Alirocumab 75 mg/ Up 150 mg Q2W
Drug: Statin — Atorvastatin, rosuvastatin and simvastatin at stable dose in participants with stable statin therapy

SUMMARY:
To determine the efficacy, long-term safety, and tolerability of alirocumab 300 mg every 4 weeks (Q4W), in comparison with placebo, as well as its potential as a starting regimen. The dose regimen of 75 mg every 2 weeks (Q2W), as used in other studies, was added as a calibrator.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women > age 18 or legal age of majority with elevated LDL-C
2. Patients not having adequate control of their hypercholesterolemia based on their individual level of CVD risk
3. Willing and able to comply with clinic visits and study-related procedures
4. Provided signed informed consent

Exclusion Criteria:

1. Recent (within 3 months prior to the screening visit) myocardial infarction, unstable angina leading to hospitalization, percutaneous coronary intervention (PCI), coronary artery bypass graft surgery (CABG), uncontrolled cardiac arrhythmia, stroke, transient ischemic attack, carotid revascularization, endovascular procedure or surgical intervention for peripheral vascular disease
2. Known history of positive test for human immunodeficiency virus (HIV)
3. Any clinically significant abnormality identified at the time of screening that in the judgment of the investigator or any sub-investigator would preclude safe completion of the study or constrain assessment of endpoints, such as major systemic diseases or participants with short life expectancy.
4. Participants considered by the investigator or any sub-investigator to be inappropriate for this study (e.g, geographic or social), actual or anticipated, that the investigator felt would restrict or limit the participant's participation for the duration of the study.
5. Certain laboratory findings obtained during the screening period

The information listed above is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial and not all inclusion/ exclusion criteria are listed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 803 (Actual)
Dates: Start 2013-09; Primary Completion 2014-09 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (83):
- United States (49):
  - Chandler, Arizona
  - Goodyear, Arizona
  - Carmichael, California
  - Fresno, California
  - West Hills, California
  - Wildomar, California
  - Colorado Springs, Colorado
  - Golden, Colorado
  - Boynton Beach, Florida
  - Jacksonville, Florida
  - Safety Harbor, Florida
  - Atlanta, Georgia
  - Boise, Idaho
  - Meridian, Idaho
  - Chicago, Illinois
  - Gurnee, Illinois
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Kansas City, Kansas
  - Louisville, Kentucky
  - Monroe, Louisiana
  - Auburn, Maine
  - Methuen, Massachusetts
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Rochester, New York
  - Farmville, North Carolina
  - Greensboro, North Carolina
  - Greenville, North Carolina
  - Raleigh, North Carolina
  - Wilson, North Carolina
  - Cincinnati, Ohio
  - Marion, Ohio
  - Tulsa, Oklahoma
  - Philadelphia, Pennsylvania
  - Wyomissing, Pennsylvania
  - Knoxville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Orem, Utah
  - Salt Lake City, Utah
  - South Jordan, Utah
  - Norfolk, Virginia
  - Richmond, Virginia
  - Spokane, Washington
  - Tacoma, Washington
  - Kenosha, Wisconsin
- Bulgaria (2):
  - Varna, Varna
  - Sofia
- Canada (7):
  - Victoria, British Columbia
  - Oshawa, Ontario
  - Toronto, Ontario
  - Woodstock, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Trois-Rivières, Quebec
- Hungary (6):
  - Budapest, Becsi Ut
  - Debrecen, HBM
  - Nyíregyháza, Sz-sz-b_m
  - Ajka, VeszprÃ©m
  - Nagykanizsa, Zala County
  - Zalaegerszeg, Zala County
- Israel (5):
  - Tel Litwinsky, IL
  - Safed, ISR
  - Ofakim, South
  - Holon
  - Tel Litwinsky
- Norway (2):
  - Skedsmokorset, Akershus
  - Oslo
- Slovakia (5):
  - Svidník, Presov
  - Bratislava, SK
  - Bratislava, SR
  - Lučenec
  - PovaÅ¾skÃ¡ Bystrica
- United Kingdom (7):
  - Worton Grange, Reading, Berkshire
  - Edgbaston, Birmingham
  - Llanishen, Cardiff
  - Choley, Lancashire
  - Waterloo, Liverpool
  - Lloyd Street North, Manchester
  - Glasgow, Scotland

REFERENCES:
- [Derived] Roth EM, Kastelein JJP, Cannon CP, Farnier M, McKenney JM, DiCioccio AT, Brunet A, Manvelian G, Sasiela WJ, Baccara-Dinet MT, Zhao J, Robinson JG. Pharmacodynamic relationship between PCSK9, alirocumab, and LDL-C lowering in the ODYSSEY CHOICE I trial. J Clin Lipidol. 2020 Sep-Oct;14(5):707-719. doi: 10.1016/j.jacl.2020.07.009. Epub 2020 Jul 25. PMID 32928709
- [Derived] Muller-Wieland D, Rader DJ, Moriarty PM, Bergeron J, Langslet G, Ray KK, Manvelian G, Thompson D, Bujas-Bobanovic M, Roth EM. Efficacy and Safety of Alirocumab 300 mg Every 4 Weeks in Individuals With Type 2 Diabetes on Maximally Tolerated Statin. J Clin Endocrinol Metab. 2019 Nov 1;104(11):5253-5262. doi: 10.1210/jc.2018-02703. PMID 31166599
- [Derived] Roth EM, Moriarty PM, Bergeron J, Langslet G, Manvelian G, Zhao J, Baccara-Dinet MT, Rader DJ; ODYSSEY CHOICE I investigators. A phase III randomized trial evaluating alirocumab 300 mg every 4 weeks as monotherapy or add-on to statin: ODYSSEY CHOICE I. Atherosclerosis. 2016 Nov;254:254-262. doi: 10.1016/j.atherosclerosis.2016.08.043. Epub 2016 Aug 31. PMID 27639753

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 97 sites in 8 countries. A total of 1491 subjects were screened between September 2013 and April 2014, 688 of whom were screen failures. Screen failures were mainly due to inclusion criteria not met.
Pre-assignment Details: Randomization was stratified according to statin therapy (with/ without) and cardiovascular risk (moderate vs. high/ very high) within the population receiving concomitant statin. Assignment to treatment arms was done using an Interactive Voice/Web Response System in 2:1:4 (Placebo: 75 mg: 300 mg) ratio after confirmation of selection criteria.
Groups:
- Placebo Q2W With Concomitant Statin: Two Subcutaneous (SC) injections of placebo (for alirocumab) every two weeks (Q2W) with stable statin therapy for 48 weeks.
- Alirocumab 75 mg Q2W/Up 150 mg Q2W With Concomitant Statin: One SC injection of each Alirocumab 75 mg and placebo Q2W with stable statin therapy for 48 weeks. Alirocumab dose up-titrated to 150 mg every two weeks (Q2W) from Week 12 when LDL-C levels ≥ 70 mg/dL (1.81 mmol/L) (for very high CV risk subjects) or ≥ 100 mg/dL (2.59 mmol/L) (for moderate and high CV risk subjects) at Week 8.
- Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin: Two SC injections of Alirocumab 150 mg every 4 weeks (Q4W) alternating with two SC injections of placebo Q4W with stable statin therapy for 48 weeks. Alirocumab dose up-titrated to 150 mg every two weeks (Q2W) from Week 12 when LDL-C levels ≥ 70 mg/dL (1.81 mmol/L) (for very high CV risk subjects) or ≥ 100 mg/dL (2.59 mmol/L) (for moderate and high CV risk subjects) at Week 8.
- Placebo Q2W Without Concomitant Statin: Two Subcutaneous (SC) injections of placebo (for alirocumab) every two weeks (Q2W) without stable statin therapy for 48 weeks.
- Alirocumab 75 mg Q2W/Up 150 mg Q2W Without Concomitant Statin: One SC injection of each Alirocumab 75 mg and placebo Q2W without stable statin therapy for 48 weeks. Alirocumab dose up-titrated to 150 mg every two weeks (Q2W) from Week 12 when LDL-C levels ≥ 70 mg/dL (1.81 mmol/L) (for very high CV risk subjects) or ≥ 100 mg/dL (2.59 mmol/L) (for moderate and high CV risk subjects) at Week 8.
- Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin: Two SC injections of Alirocumab 150 mg every 4 weeks (Q4W) alternating with two SC injections of placebo Q4W without stable statin therapy for 48 weeks. Alirocumab dose up-titrated to 150 mg every two weeks (Q2W) from Week 12 when LDL-C levels ≥ 70 mg/dL (1.81 mmol/L) (for very high CV risk subjects) or ≥ 100 mg/dL (2.59 mmol/L) (for moderate and high CV risk subjects) at Week 8.
Period: Overall Study
Arm/Group | Placebo Q2W With Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W With Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin | Placebo Q2W Without Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W Without Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin
Started | 157 | 78 | 312 | 73 | 37 | 146
Treated | 157 | 78 | 312 | 72 | 37 | 146
Completed 24 Weeks Treatment Period | 137 | 68 | 285 | 58 | 31 | 120
Completed | 129 | 65 | 272 | 53 | 29 | 105
Not Completed | 28 | 13 | 40 | 20 | 8 | 41
Not completed — Participant moved | 2 | 0 | 1 | 1 | 0 | 3
Not completed — Physician Decision | 0 | 2 | 1 | 1 | 0 | 0
Not completed — Other than specified | 2 | 3 | 5 | 12 | 4 | 11
Not completed — Adverse Event | 13 | 4 | 17 | 4 | 3 | 14
Not completed — Poor compliance to protocol | 5 | 3 | 8 | 0 | 1 | 6
Not completed — Randomized and not treated | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 1 | 8 | 1 | 0 | 5
Not completed — Related to study drug administration | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All randomized population regardless of concomitant statin therapy.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Q2W With Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W With Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin | Placebo Q2W Without Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W Without Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin | Total
Number analyzed (Participants) | 157 | 78 | 312 | 73 | 37 | 146 | 803
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (9.7) | 60.7 (9.1) | 61.6 (10) | 59.4 (10.2) | 59.3 (11.3) | 59.2 (10.8) | 60.8 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 27 | 122 | 33 | 23 | 80 | 341
  Male | 101 | 51 | 190 | 40 | 14 | 66 | 462
Calculated LDL-C in mg/dL [Mean (Standard Deviation); unit: mg/dL] — Calculated LDL-C from Friedewald formula (LDL-C = Total cholesterol - High-density lipoprotein cholesterol - [Triglyceride/5])
  mg/dL | 112.1 (37.3) | 114.9 (36) | 112.4 (32.8) | 131 (30.4) | 148.4 (36.8) | 146.1 (33.5) | 122.1 (36.9)
Calculated LDL-C in mmol/L [Mean (Standard Deviation); unit: mmol/L] | 2.903 (0.965) | 2.977 (0.933) | 2.912 (0.85) | 3.392 (0.787) | 3.842 (0.953) | 3.785 (0.868) | 3.162 (0.956)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Calculated LDL-C in Participants Not Receiving Concomitant Statin Therapy - ITT Analysis
Description: Adjusted LS means and standard errors at Week 24 and at averaged Week 21 to 24 from MMRM including available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment. ITT population (subjects without concomitant statin therapy): all randomized subjects who did not receive concomitant statin therapy, with one baseline and at least one post-baseline calculated LDL-C value on- or off-treatment. Alirocumab 75 mg Q2W arm (calibrator arm) was included only to facilitate comparison of results of this study with the results of other studies that used an alirocumab 75 mg Q2W regimen. Hence no statistical comparison was performed for this arm.
Time Frame: From Baseline to Week 24
Population: ITT population (participants without concomitant statin therapy): all randomized participants who did not receive concomitant statin therapy, with one baseline and at least one post-baseline calculated LDL-C value on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W Without Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W Without Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin
Number analyzed (Participants) | 71 | 37 | 144
percent change
  At Week 24 | -0.3 (2.7) | -50.2 (3.7) | -52.7 (1.9)
  At averaged Week 21 to 24 | -1.6 (2.6) | -54 (3.6) | -56.9 (1.8)
Statistical Analysis 1: Comparison: Placebo Q2W Without Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin; At Week 24; Test type: Superiority or Other — Alirocumab 300 mg group was compared to placebo group using an appropriate contrast statement; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.025; LS Mean Difference = -52.4, 97.5% CI 2-sided [-59.8 to -45.0]
Statistical Analysis 2: Comparison: Placebo Q2W Without Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin; Week 21-24; Test type: Superiority or Other — Alirocumab 300 mg group was compared to placebo group using an appropriate contrast statement; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.025; LS Mean Difference = -55.2, 97.5% CI 2-sided [-62.3 to -48.1]

2. Primary Outcome: Percent Change From Baseline in Calculated LDL-C in Participants Receiving Concomitant Statin Therapy - Intent-to-Treat (ITT Analysis)
Description: Adjusted least squares (LS) means and standard errors at Week 24 and at averaged Week 21 to 24 were obtained from a mixed effect model with repeated measures (MMRM) model to account for missing data. All available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment were used in this model (ITT analysis). ITT population (subjects with concomitant statin therapy): all randomized subjects who received concomitant statin therapy, with one baseline and at least one post-baseline calculated LDL-C value on- or off-treatment. Alirocumab 75 mg Q2W arm (calibrator arm) was included only to facilitate comparison of results of this study with the results of other studies that used an alirocumab 75 mg Q2W regimen. Hence no statistical comparison was performed for this arm.
Time Frame: From Baseline to Week 24
Population: ITT population (participants with concomitant statin therapy): all randomized participants who received concomitant statin therapy, with one baseline and at least one post-baseline calculated LDL-C value on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W With Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W With Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin
Number analyzed (Participants) | 156 | 76 | 308
percent change
  At Week 24 | -0.1 (2.3) | -51.6 (3.3) | -58.8 (1.6)
  At averaged Week 21 to 24 | 0.8 (2.0) | -57.9 (2.8) | -65.8 (1.4)
Statistical Analysis 1: Comparison: Placebo Q2W With Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin; At Week 24; Test type: Superiority or Other — Alirocumab 300 mg group was compared to placebo group using an appropriate contrast statement; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.025; LS Mean Difference = -58.7, 97.5% CI 2-sided [-65.0 to -52.4]
Statistical Analysis 2: Comparison: Placebo Q2W With Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin; Week 21-24; Test type: Superiority or Other — Alirocumab 300 mg group was compared to placebo group using an appropriate contrast statement; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.025; LS Mean Difference = -65, 97.5% CI 2-sided [-70.4 to -59.5]

3. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 24 in Participants Not Receiving Concomitant Statin Therapy - On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 24 were obtained from MMRM model including available post-baseline on-treatment data from Week 4 to Week 24 (i.e. up to 21 days after last injection) (on-treatment analysis). Modified ITT (mITT) population (subjects with or without concomitant statin therapy): all randomized and treated subjects who did not receive concomitant statin therapy, with one baseline and at least one post-baseline calculated LDL-C value on-treatment. Alirocumab 75 mg Q2W arm (calibrator arm) was included only to facilitate comparison of results of this study with the results of other studies that used an alirocumab 75 mg Q2W regimen. Hence no statistical comparison was performed for this arm.
Time Frame: From Baseline to Week 24
Population: Modified ITT (mITT) population (participants without concomitant statin therapy): all randomized and treated participants who did not receive concomitant statin therapy, with one baseline and at least one post-baseline calculated LDL-C value on-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W Without Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W Without Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin
Number analyzed (Participants) | 70 | 37 | 141
percent change | -0.4 (2.0) | -54.6 (2.8) | -59.4 (1.4)
Statistical Analysis 1: Comparison: Placebo Q2W Without Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin; A hierarchical testing procedure was used to control type I error and handle multiple secondary endpoint analyses. Testing was then performed sequentially in the order the endpoints are reported. The hierarchical testing sequence continued only when previous endpoint was statistically significant at 0.025 level; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.025; LS Mean Difference = -59.0, 97.5% CI 2-sided [-64.6 to -53.4]

4. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 24 in Participants Receiving Concomitant Statin Therapy - On-Treatment Analysis
Description: as for outcome 3
Time Frame: From Baseline to Week 24
Population: mITT population
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W With Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W With Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin
Number analyzed (Participants) | 151 | 75 | 302
percent change | -0.3 (2.1) | -55.1 (3.0) | -62.3 (1.5)
Statistical Analysis 1: Comparison: Placebo Q2W With Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.025; LS Mean Difference = -62.0, 97.5% CI 2-sided [-67.7 to -56.2]

5. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 12 in Participants Not Receiving Concomitant Statin Therapy - ITT Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM model including available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment. ITT population (subjects with or without concomitant statin therapy). Alirocumab 75 mg Q2W arm (calibrator arm) was included only to facilitate comparison of results of this study with the results of other studies that used an alirocumab 75 mg Q2W regimen. Hence no statistical comparison was performed for this arm.
Time Frame: From Baseline to Week 12
Population: ITT population (participants without concomitant statin therapy)
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W Without Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W Without Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin
Number analyzed (Participants) | 71 | 37 | 144
percent change | 0.3 (2.1) | -51.8 (2.9) | -58.4 (1.4)
Statistical Analysis 1: Comparison: Placebo Q2W Without Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.025; LS Mean Difference = -58.7, 97.5% CI 2-sided [-64.5 to -53.0]

6. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 12 in Participants Receiving Concomitant Statin Therapy - ITT Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 12
Population: ITT population (participants with concomitant statin therapy)
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W With Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W With Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin
Number analyzed (Participants) | 156 | 76 | 308
percent change | 1.1 (2.2) | -45.3 (3.1) | -55.3 (1.5)
Statistical Analysis 1: Comparison: Placebo Q2W With Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.025; LS Mean Difference = -56.3, 97.5% CI 2-sided [-62.3 to -50.3]

7. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 12 in Participants Not Receiving Concomitant Statin Therapy - On-treatment Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 12
Population: mITT population (participants without concomitant statin therapy)
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W Without Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W Without Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin
Number analyzed (Participants) | 70 | 37 | 141
percent change | -0.5 (2.0) | -53.9 (2.7) | -60.0 (1.4)
Statistical Analysis 1: Comparison: Placebo Q2W Without Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.025; LS Mean Difference = -59.5, 97.5% CI 2-sided [-65.0 to -54.1]

8. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 12 in Participants Receiving Concomitant Statin Therapy - On-treatment Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 12
Population: mITT population (participants with concomitant statin therapy)
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W With Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W With Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin
Number analyzed (Participants) | 151 | 75 | 302
percent change | 1.4 (1.9) | -47.3 (2.8) | -58.0 (1.4)
Statistical Analysis 1: Comparison: Placebo Q2W With Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.025; LS Mean Difference = -59.4, 97.5% CI 2-sided [-64.8 to -54.0]

9. Secondary Outcome: Percent Change From Baseline in Apolipoprotein (Apo) B at Week 24 in Participants Not Receiving Concomitant Statin Therapy - ITT Analysis
Description: Adjusted LS means and standard errors at Week 24 from MMRM model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment. Subjects of the ITT population (with or without concomitant statin therapy) with one baseline and at least one post-baseline Apo B value on- or off-treatment (Apo B ITT population). Alirocumab 75 mg Q2W arm (calibrator arm) was included only to facilitate comparison of results of this study with the results of other studies that used an alirocumab 75 mg Q2W regimen. Hence no statistical comparison was performed for this arm.
Time Frame: From Baseline to Week 24
Population: Apo B ITT population (participants without concomitant statin therapy)
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W Without Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W Without Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin
Number analyzed (Participants) | 71 | 34 | 138
percent change | -0.7 (2.3) | -39.0 (3.3) | -40.2 (1.6)
Statistical Analysis 1: Comparison: Placebo Q2W Without Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.025; LS Mean Difference = -39.5, 97.5% CI 2-sided [-45.8 to -33.1]

10. Secondary Outcome: Percent Change From Baseline in Apo B at Week 24 in Participants Receiving Concomitant Statin Therapy - ITT Analysis
Description: as for outcome 9
Time Frame: From Baseline to Week 24
Population: Apo B ITT population (participants with concomitant statin therapy)
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W With Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W With Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin
Number analyzed (Participants) | 146 | 75 | 292
percent change | 3.1 (1.8) | -36.7 (2.6) | -45.1 (1.3)
Statistical Analysis 1: Comparison: Placebo Q2W With Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.025; LS Mean Difference = -48.2, 97.5% CI 2-sided [-53.2 to -43.2]

11. Secondary Outcome: Percent Change From Baseline in Apo B at Week 24 in Participants Not Receiving Concomitant Statin Therapy - On-Treatment Analysis
Description: as for outcome 9
Time Frame: From Baseline to Week 24
Population: Apo B mITT population (participants without concomitant statin therapy)
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W Without Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W Without Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin
Number analyzed (Participants) | 70 | 37 | 141
percent change | -0.3 (2.0) | -42.0 (2.7) | -44.8 (1.4)
Statistical Analysis 1: Comparison: Placebo Q2W Without Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.025; LS Mean Difference = -44.5, 97.5% CI 2-sided [-49.9 to -39.1]

12. Secondary Outcome: Percent Change From Baseline in Apo B at Week 24 in Participants Receiving Concomitant Statin Therapy - On-Treatment Analysis
Description: as for outcome 9
Time Frame: From Baseline to Week 24
Population: Apo B mITT population (participants with concomitant statin therapy)
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W With Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W With Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin
Number analyzed (Participants) | 142 | 74 | 286
percent change | 3.1 (1.7) | -38.3 (2.5) | -47.2 (1.2)
Statistical Analysis 1: Comparison: Placebo Q2W With Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.025; LS Mean Difference = -50.3, 97.5% CI 2-sided [-55.0 to -45.6]

13. Secondary Outcome: Percent Change From Baseline in Non-High Density Lipoprotein Cholesterol (Non-HDL-C) at Week 24 in Participants Not Receiving Concomitant Statin Therapy - ITT Analysis
Description: Adjusted LS means and standard errors at Week 24 from MMRM model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment. Subjects of the ITT population (with or without concomitant statin therapy) with one baseline and at least one post-baseline non-HDL-C value on- or off-treatment (non-HDL-C ITT population). Alirocumab 75 mg Q2W arm (calibrator arm) was included only to facilitate comparison of results of this study with the results of other studies that used an alirocumab 75 mg Q2W regimen. Hence no statistical comparison was performed for this arm.
Time Frame: From Baseline to Week 24
Population: Non-HDL-C ITT population (participants without concomitant statin therapy)
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W Without Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W Without Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin
Number analyzed (Participants) | 71 | 37 | 144
percent change | -0.3 (2.5) | -43.6 (3.4) | -43.3 (1.7)
Statistical Analysis 1: Comparison: Placebo Q2W Without Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.025; LS Mean Difference = -43.0, 97.5% CI 2-sided [-49.9 to -36.2]

14. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 24 in Participants Receiving Concomitant Statin Therapy - ITT Analysis
Description: as for outcome 13
Time Frame: From Baseline to Week 24
Population: Non-HDL-C ITT population (participants with concomitant statin therapy)
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W With Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W With Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin
Number analyzed (Participants) | 156 | 76 | 308
percent change | 0.3 (1.9) | -41.6 (2.7) | -49.7 (1.3)
Statistical Analysis 1: Comparison: Placebo Q2W With Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.025; LS Mean Difference = -50.0, 97.5% CI 2-sided [-55.3 to -44.8]

15. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 24 in Participants Not Receiving Concomitant Statin Therapy - On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 24 from MMRM model including available post-baseline on-treatment data from Week 4 to Week 24 (i.e. up to 21 days after last injection). Subjects of the mITT population (with or without concomitant statin therapy) with one baseline and at least one post-baseline non-HDL-C value on-treatment (non-HDL-C mITT population). Alirocumab 75 mg Q2W arm (calibrator arm) was included only to facilitate comparison of results of this study with the results of other studies that used an alirocumab 75 mg Q2W regimen. Hence no statistical comparison was performed for this arm.
Time Frame: From Baseline to Week 24
Population: Non-HDL-C mITT population (participants without concomitant statin therapy)
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W Without Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W Without Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin
Number analyzed (Participants) | 70 | 37 | 141
percent change | 0.1 (2.1) | -47.2 (2.8) | -48.9 (1.4)
Statistical Analysis 1: Comparison: Placebo Q2W Without Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.025; LS Mean Difference = -49.0, 97.5% CI 2-sided [-54.8 to -43.3]

16. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 24 in Participants Receiving Concomitant Statin Therapy - On-Treatment Analysis
Description: as for outcome 15
Time Frame: From Baseline to Week 24
Population: Non-HDL-C mITT population (participants with concomitant statin therapy)
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W With Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W With Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin
Number analyzed (Participants) | 151 | 75 | 302
percent change | 0.2 (1.8) | -44.4 (2.5) | -52.6 (1.2)
Statistical Analysis 1: Comparison: Placebo Q2W With Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.025; LS Mean Difference = -52.8, 97.5% CI 2-sided [-57.6 to -47.9]

17. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (Total-C) at Week 24 in Participants Not Receiving Concomitant Statin Therapy - ITT Analysis
Description: Adjusted LS means and standard errors at Week 24 from MMRM model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment. Subjects of the ITT population (with or without concomitant statin therapy) with one baseline and at least one post-baseline Total-C value on- or off-treatment (Total-C ITT population). Alirocumab 75 mg Q2W arm (calibrator arm) was included only to facilitate comparison of results of this study with the results of other studies that used an alirocumab 75 mg Q2W regimen. Hence no statistical comparison was performed for this arm.
Time Frame: From Baseline to Week 24
Population: Total-C ITT population (participants without concomitant statin therapy)
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W Without Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W Without Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin
Number analyzed (Participants) | 71 | 37 | 144
percent change | -1.9 (1.9) | -32.5 (2.6) | -33.3 (1.3)
Statistical Analysis 1: Comparison: Placebo Q2W Without Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.025; LS Mean Difference = -31.4, 97.5% CI 2-sided [-36.6 to -26.3]

18. Secondary Outcome: Percent Change From Baseline in Total-C at Week 24 in Participants Receiving Concomitant Statin Therapy - ITT Analysis
Description: as for outcome 17
Time Frame: From Baseline to Week 24
Population: Total-C ITT population (participants with concomitant statin therapy)
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W With Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W With Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin
Number analyzed (Participants) | 156 | 76 | 308
percent change | -0.8 (1.4) | -30.0 (2.0) | -35.8 (1.0)
Statistical Analysis 1: Comparison: Placebo Q2W With Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.025; LS Mean Difference = -35.0, 97.5% CI 2-sided [-38.9 to -31.1]

19. Secondary Outcome: Percent Change From Baseline in Apo B at Week 12 in Participants Not Receiving Concomitant Statin Therapy - ITT Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment. Apo B ITT population (subjects with or without concomitant statin therapy). Alirocumab 75 mg Q2W arm (calibrator arm) was included only to facilitate comparison of results of this study with the results of other studies that used an alirocumab 75 mg Q2W regimen. Hence no statistical comparison was performed for this arm.
Time Frame: From Baseline to Week 12
Population: Apo B ITT population (participants without concomitant statin therapy)
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W Without Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W Without Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin
Number analyzed (Participants) | 71 | 34 | 138
percent change | -2.3 (1.7) | -40.8 (2.5) | -46.4 (1.3)
Statistical Analysis 1: Comparison: Placebo Q2W Without Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.025; LS Mean Difference = -44.1, 97.5% CI 2-sided [-49.0 to -39.2]

20. Secondary Outcome: Percent Change From Baseline in Apo B at Week 12 in Participants Receiving Concomitant Statin Therapy - ITT Analysis
Description: as for outcome 19
Time Frame: From Baseline to Week 12
Population: Apo B ITT population (participants with concomitant statin therapy).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W With Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W With Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin
Number analyzed (Participants) | 146 | 75 | 292
percent change | 3.6 (1.8) | -33.0 (2.5) | -41.2 (1.3)
Statistical Analysis 1: Comparison: Placebo Q2W With Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.025; LS Mean Difference = -44.8, 97.5% CI 2-sided [-49.7 to -39.9]

21. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 12 in Participants Not Receiving Concomitant Statin Therapy - ITT Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment. Non-HDL-C ITT population (subjects with or without concomitant statin therapy). Alirocumab 75 mg Q2W arm (calibrator arm) was included only to facilitate comparison of results of this study with the results of other studies that used an alirocumab 75 mg Q2W regimen. Hence no statistical comparison was performed for this arm.
Time Frame: From Baseline to Week 12
Population: Non-HDL-C ITT population (participants without concomitant statin therapy).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W Without Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W Without Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin
Number analyzed (Participants) | 71 | 37 | 144
percent change | -0.4 (1.8) | -45.8 (2.5) | -49.9 (1.3)
Statistical Analysis 1: Comparison: Placebo Q2W Without Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.025; LS Mean Difference = -49.5, 97.5% CI 2-sided [-54.5 to -44.6]

22. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 12 in Participants Receiving Concomitant Statin Therapy - ITT Analysis
Description: as for outcome 21
Time Frame: From Baseline to Week 12
Population: Non-HDL-C ITT population (participants with concomitant statin therapy).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W With Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W With Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin
Number analyzed (Participants) | 156 | 76 | 308
percent change | 0.6 (1.9) | -37.4 (2.7) | -46.5 (1.3)
Statistical Analysis 1: Comparison: Placebo Q2W With Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.025; LS Mean Difference = -47.1, 97.5% CI 2-sided [-52.2 to -42.0]

23. Secondary Outcome: Percent Change From Baseline in Total-C at Week 12 in Participants Not Receiving Concomitant Statin Therapy - ITT Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment. Total-C ITT population (subjects with or without concomitant statin therapy). Alirocumab 75 mg Q2W arm (calibrator arm) was included only to facilitate comparison of results of this study with the results of other studies that used an alirocumab 75 mg Q2W regimen. Hence no statistical comparison was performed for this arm.
Time Frame: From Baseline to Week 12
Population: Total-C ITT population (participants without concomitant statin therapy)
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W Without Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W Without Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin
Number analyzed (Participants) | 71 | 37 | 144
percent change | -1.0 (1.4) | -33.4 (2.0) | -37.4 (1.0)
Statistical Analysis 1: Comparison: Placebo Q2W Without Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.025; LS Mean Difference = -36.4, 97.5% CI 2-sided [-40.4 to -32.4]

24. Secondary Outcome: Percent Change From Baseline in Total-C at Week 12 in Participants Receiving Concomitant Statin Therapy - ITT Analysis
Description: as for outcome 23
Time Frame: From Baseline to Week 12
Population: Total-C ITT population (participants with concomitant statin therapy)
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W With Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W With Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin
Number analyzed (Participants) | 156 | 76 | 308
percent change | -0.1 (1.3) | -26.5 (1.9) | -32.9 (1.0)
Statistical Analysis 1: Comparison: Placebo Q2W With Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.025; LS Mean Difference = -32.8, 97.5% CI 2-sided [-36.5 to -29.1]

25. Secondary Outcome: Percentage of Very High CV Risk Participants Reaching Calculated LDL-C<70 mg/dL or Moderate or High CV Risk Participants Reaching Calculated LDL-C<100 mg/dL (Without Concomitant Statin Therapy) at Week 24 - ITT Analysis
Description: Very high CV risk: history of documented coronary heart disease (CHD) or CHD risk equivalent. High CV risk: calculated 10-year fatal CVD risk score ≥5%, moderate chronic kidney disease, type 1/type 2 diabetes mellitus (DM) without target organ damage, or heFH not meeting definition of very high risk. Moderate CV risk: calculated 10-year fatal CVD risk score ≥1 &<5%. CHD risk equivalent: peripheral arterial disease, ischemic stroke, transient ischemic attack, abdominal aortic aneurysm, carotid artery(CA)occlusion>50%, carotid endarterectomy/CA stent procedure, renal artery stenosis/stent procedure, type 1/type 2 DM with target organ damage. Adjusted percentages at Week 24 obtained from multiple imputation approach model for handling of missing data. All available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment included in imputation model. ITT population (subjects with or without concomitant statin therapy).
Time Frame: Up to Week 24
Population: ITT population (participants without concomitant statin therapy)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W Without Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W Without Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin
Number analyzed (Participants) | 71 | 37 | 144
percentage of participants | 9.4 | 84.9 | 78.9
Statistical Analysis 1: Comparison: Placebo Q2W Without Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant). Statistical analysis used a multiple imputation approach followed by logistic regression model; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.025; Multiple imputation approach followed by logistic regression model; Odds Ratio (OR) = 68.0, 97.5% CI 2-sided [20.9 to 221.0]

26. Secondary Outcome: Percentage of Very High Cardiovascular (CV) Risk Participants Reaching Calculated LDL-C <70 mg/dL or Moderate or High CV Risk Participants Reaching Calculated LDL-C <100 mg/dL (With Concomitant Statin Therapy) at Week 24 - ITT Analysis
Description: as for outcome 25
Time Frame: Up to Week 24
Population: ITT population (participants with concomitant statin therapy)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W With Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W With Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin
Number analyzed (Participants) | 156 | 76 | 308
percentage of participants | 22.2 | 82.5 | 85.2
Statistical Analysis 1: Comparison: Placebo Q2W With Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant). Statistical analysis used multiple imputation approach followed by logistic regression model; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.025; Odds Ratio (OR) = 25.6, 97.5% CI 2-sided [13.7 to 47.8]

27. Secondary Outcome: Percentage of Very High CV Risk Participants Reaching Calculated LDL-C<70 mg/dL (1.81 mmol/L) or Moderate or High CV Risk Participants Reaching Calculated LDL-C<100 mg/dL(2.59 mmol/L) (Without Concomitant Statin Therapy) at Week 24 - On-Treatment Analysis
Description: Adjusted percentages at Week 24 were from multiple imputation approach model including available post-baseline on-treatment data from Week 4 to Week 24 (i.e. up to 21 days after last injection). mITT population (subjects with or without concomitant statin therapy). Alirocumab 75 mg Q2W arm (calibrator arm) was included only to facilitate comparison of results of this study with the results of other studies that used an alirocumab 75 mg Q2W regimen. Hence no statistical comparison was performed for this arm.
Time Frame: Up to Week 24
Population: mITT population (participants without concomitant statin therapy)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W Without Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W Without Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin
Number analyzed (Participants) | 70 | 37 | 141
percentage of participants | 11.3 | 93.0 | 88.6
Statistical Analysis 1: Comparison: Placebo Q2W Without Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.025; Multiple imputation approach followed by logistic regression model; Odds Ratio (OR) = 280.2, 97.5% CI 2-sided [56.7 to 1385.7]

28. Secondary Outcome: Percentage of Very High CV Risk Participants Reaching Calculated LDL-C <70 mg/dL(1.81 mmol/L) or Moderate or High CV Risk Participants Reaching Calculated LDL-C <100 mg/dL(2.59 mmol/L) (With Concomitant Statin Therapy) at Week 24 - On-Treatment Analysis
Description: as for outcome 27
Time Frame: Up to Week 24
Population: mITT population (participants with concomitant statin therapy)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W With Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W With Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin
Number analyzed (Participants) | 151 | 75 | 302
percentage of participants | 22.5 | 86.4 | 89.5
Statistical Analysis 1: Comparison: Placebo Q2W With Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin; [analysis description as in outcome 25, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.025; Odds Ratio (OR) = 41.3, 97.5% CI 2-sided [20.3 to 83.8]

29. Secondary Outcome: Percentage of Participants (Without Concomitant Statin Therapy) Reaching Calculated LDL-C <70 mg/dL (1.81 mmol/L) at Week 24 - ITT Analysis
Description: Adjusted percentages at Week 24 were obtained from multiple imputation approach model for handling of missing data. All available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment were included in the imputation model. ITT population (subjects with or without concomitant statin therapy). Alirocumab 75 mg Q2W arm (calibrator arm) was included only to facilitate comparison of results of this study with the results of other studies that used an alirocumab 75 mg Q2W regimen. Hence no statistical comparison was performed for this arm.
Time Frame: Up to Week 24
Population: ITT population (participants without concomitant statin therapy)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W Without Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W Without Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin
Number analyzed (Participants) | 71 | 37 | 144
percentage of participants | 3.3 | 57.7 | 62.0
Statistical Analysis 1: Comparison: Placebo Q2W Without Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin; [analysis description as in outcome 25, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.025; Odds Ratio (OR) = 90.6, 97.5% CI 2-sided [16.5 to 498.3]

30. Secondary Outcome: Percentage of Participants (With Concomitant Statin Therapy) Reaching Calculated LDL-C <70 mg/dL (1.81 mmol/L) at Week 24 - ITT Analysis
Description: as for outcome 29
Time Frame: Up to Week 24
Population: ITT population (participants with concomitant statin therapy)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W With Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W With Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin
Number analyzed (Participants) | 156 | 76 | 308
percentage of participants | 10.9 | 74.4 | 80.4
Statistical Analysis 1: Comparison: Placebo Q2W With Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin; [analysis description as in outcome 25, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.025; Odds Ratio (OR) = 49.5, 97.5% CI 2-sided [23.4 to 104.4]

31. Secondary Outcome: Percentage of Participants (Without Concomitant Statin Therapy) Reaching Calculated LDL-C <70 mg/dL (1.81 mmol/L) at Week 24 - On-Treatment Analysis
Description: Adjusted percentages at Week 24 from multiple imputation approach model including available post-baseline data from Week 4 to Week 24 (i.e. up to 21 days after last injection). mITT population (subjects with or without concomitant statin therapy). Alirocumab 75 mg Q2W arm (calibrator arm) was included only to facilitate comparison of results of this study with the results of other studies that used an alirocumab 75 mg Q2W regimen. Hence no statistical comparison was performed for this arm.
Time Frame: Up to Week 24
Population: mITT population (participants without concomitant statin therapy)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W Without Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W Without Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin
Number analyzed (Participants) | 70 | 37 | 141
percentage of participants | 2.1 | 61.7 | 70.4
Statistical Analysis 1: Comparison: Placebo Q2W Without Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin; [analysis description as in outcome 26, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.025; Odds Ratio (OR) = 297.1, 97.5% CI 2-sided [27.9 to 3160.6]

32. Secondary Outcome: Percentage of Participants (With Concomitant Statin Therapy) Reaching Calculated LDL-C <70 mg/dL (1.81 mmol/L) at Week 24 - On-Treatment Analysis
Description: as for outcome 31
Time Frame: Up to Week 24
Population: mITT population (participants with concomitant statin therapy)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W With Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W With Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin
Number analyzed (Participants) | 151 | 75 | 302
percentage of participants | 10.8 | 77.4 | 84.8
Statistical Analysis 1: Comparison: Placebo Q2W With Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin; [analysis description as in outcome 26, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.025; Odds Ratio (OR) = 77.7, 97.5% CI 2-sided [34.1 to 176.8]

33. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a) in Participants Not Receiving Concomitant Statin Therapy at Week 24 - ITT Analysis
Description: Adjusted means and standard errors at Week 24 from a multiple imputation approach followed by robust regression model for handling of missing data. All available post-baseline data from Week 4 to Week 24 regardless of status on-or off-treatment were included in the imputation model. ITT population (subjects with or without concomitant statin therapy). Alirocumab 75 mg Q2W arm (calibrator arm) was included only to facilitate comparison of results of this study with the results of other studies that used an alirocumab 75 mg Q2W regimen. Hence no statistical comparison was performed for this arm.
Time Frame: From Baseline to Week 24
Population: ITT population (participants without concomitant statin therapy)
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W Without Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W Without Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin
Number analyzed (Participants) | 71 | 37 | 144
percent change | 6.4 (3.4) | -14.0 (4.8) | -21.3 (2.4)
Statistical Analysis 1: Comparison: Placebo Q2W Without Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant). Statistical analysis used a multiple imputation approach followed by a robust regression model; Test type: Superiority or Other; p < 0.0001, Regression, Robust — Threshold for significance ≤ 0.025; Adjusted Mean Difference = -27.7, 97.5% CI 2-sided [-37.0 to -18.3]

34. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a) in Participants Receiving Concomitant Statin Therapy at Week 24 - ITT Analysis
Description: as for outcome 33
Time Frame: From Baseline to Week 24
Population: ITT population (participants with concomitant statin therapy)
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W With Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W With Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin
Number analyzed (Participants) | 156 | 76 | 308
percent change | 9.8 (2.4) | -16.9 (3.3) | -19.3 (1.6)
Statistical Analysis 1: Comparison: Placebo Q2W With Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin; [analysis description as in outcome 33, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Robust — Threshold for significance ≤ 0.025; Adjusted Mean Difference = -29.1, 97.5% CI 2-sided [-35.5 to -22.7]

35. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a) in Participants Not Receiving Concomitant Statin Therapy at Week 12 - ITT Analysis
Description: Adjusted means and standard errors at Week 12 from multiple imputation approach followed by robust regression model including all available post-baseline data from Week 4 to Week 24 regardless of status on-or off-treatment. ITT population (subjects with or without concomitant statin therapy). Alirocumab 75 mg Q2W arm (calibrator arm) was included only to facilitate comparison of results of this study with the results of other studies that used an alirocumab 75 mg Q2W regimen. Hence no statistical comparison was performed for this arm.
Time Frame: From Baseline to Week 12
Population: ITT population (participants without concomitant statin therapy)
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W Without Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W Without Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin
Number analyzed (Participants) | 71 | 37 | 144
percent change | -5.5 (3.3) | -26.9 (4.7) | -28.9 (2.3)
Statistical Analysis 1: Comparison: Placebo Q2W Without Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin; [analysis description as in outcome 33, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Robust — Threshold for significance ≤ 0.025; Adjusted Mean Difference = -23.5, 97.5% CI 2-sided [-32.4 to -14.5]

36. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a) in Participants Receiving Concomitant Statin Therapy at Week 12 - ITT Analysis
Description: as for outcome 35
Time Frame: From Baseline to Week 12
Population: ITT population (participants with concomitant statin therapy)
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W With Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W With Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin
Number analyzed (Participants) | 156 | 76 | 308
percent change | 7.0 (2.3) | -12.4 (3.2) | -19.6 (1.6)
Statistical Analysis 1: Comparison: Placebo Q2W With Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin; [analysis description as in outcome 33, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Robust — Threshold for significance ≤ 0.025; Adjusted Mean Difference = -26.6, 97.5% CI 2-sided [-32.8 to -20.4]

37. Secondary Outcome: Percent Change From Baseline in HDL-C in Participants Not Receiving Concomitant Statin Therapy at Week 24 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 24 from MMRM model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment. Subjects of the ITT population (with or without concomitant statin therapy) with one baseline and at least one post-baseline HDL-C value on- or off-treatment (HDL-C ITT population). Alirocumab 75 mg Q2W arm (calibrator arm) was included only to facilitate comparison of results of this study with the results of other studies that used an alirocumab 75 mg Q2W regimen. Hence no statistical comparison was performed for this arm.
Time Frame: From Baseline to Week 24
Population: HDL-C ITT population (participants without concomitant statin therapy)
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W Without Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W Without Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin
Number analyzed (Participants) | 71 | 37 | 144
percent change | -5.3 (1.7) | -0.1 (2.4) | 2.5 (1.2)
Statistical Analysis 1: Comparison: Placebo Q2W Without Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis — Threshold for significance ≤ 0.025; LS Mean Difference = 7.8, 97.5% CI 2-sided [3.1 to 12.6]

38. Secondary Outcome: Percent Change From Baseline in HDL-C in Participants Receiving Concomitant Statin Therapy at Week 24 - ITT Analysis
Description: as for outcome 37
Time Frame: From Baseline to Week 24
Population: HDL-C ITT population (participants with concomitant statin therapy)
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W With Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W With Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin
Number analyzed (Participants) | 156 | 76 | 308
percent change | -1.5 (1.2) | 6.0 (1.7) | 3.6 (0.8)
Statistical Analysis 1: Comparison: Placebo Q2W With Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis — Threshold for significance ≤ 0.025; LS Mean Difference = 5.1, 97.5% CI 2-sided [1.9 to 8.4]

39. Secondary Outcome: Percent Change From Baseline in HDL-C in Participants Not Receiving Concomitant Statin Therapy at Week 12 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment. HDL-C ITT population (subjects with or without concomitant statin therapy). Alirocumab 75 mg Q2W arm (calibrator arm) was included only to facilitate comparison of results of this study with the results of other studies that used an alirocumab 75 mg Q2W regimen. Hence no statistical comparison was performed for this arm.
Time Frame: From Baseline to Week 12
Population: HDL-C ITT population (participants without concomitant statin therapy)
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W Without Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W Without Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin
Number analyzed (Participants) | 71 | 37 | 144
percent change | -0.9 (1.6) | 2.5 (2.2) | 6.0 (1.1)
Statistical Analysis 1: Comparison: Placebo Q2W Without Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis — Threshold for significance ≤ 0.025; LS Mean Difference = 6.9, 97.5% CI 2-sided [2.6 to 11.1]

40. Secondary Outcome: Percent Change From Baseline in HDL-C in Participants Receiving Concomitant Statin Therapy at Week 12 - ITT Analysis
Description: as for outcome 39
Time Frame: From Baseline to Week 12
Population: HDL-C ITT population (participants with concomitant statin therapy)
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W With Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W With Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin
Number analyzed (Participants) | 156 | 76 | 308
percent change | 0.4 (1.2) | 7.6 (1.8) | 5.7 (0.9)
Statistical Analysis 1: Comparison: Placebo Q2W With Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0007, Mixed Models Analysis — Threshold for significance ≤ 0.025; LS Mean Difference = 5.2, 97.5% CI 2-sided [1.8 to 8.7]

41. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides in Participants Not Receiving Concomitant Statin Therapy at Week 24 - ITT Analysis
Description: Adjusted means and standard errors at Week 24 from multiple imputation approach followed by robust regression model including all available post-baseline data from Week 4 to Week 24 regardless of status on-or off-treatment. ITT population (subjects with or without concomitant statin therapy). Alirocumab 75 mg Q2W arm (calibrator arm) was included only to facilitate comparison of results of this study with the results of other studies that used an alirocumab 75 mg Q2W regimen. Hence no statistical comparison was performed for this arm.
Time Frame: From Baseline to Week 24
Population: ITT population (participants without concomitant statin therapy)
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W Without Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W Without Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin
Number analyzed (Participants) | 71 | 37 | 144
percent change | -1.5 (3.4) | -9.8 (4.9) | -13.4 (2.5)
Statistical Analysis 1: Comparison: Placebo Q2W Without Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin; [analysis description as in outcome 33, analysis 1]; Test type: Superiority or Other; p = 0.0042, Regression, Robust — Threshold for significance ≤ 0.025; Adjusted Mean Difference = -11.9, 97.5% CI 2-sided [-21.3 to -2.6]

42. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides in Participants Receiving Concomitant Statin Therapy at Week 24 - ITT Analysis
Description: as for outcome 41
Time Frame: From Baseline to Week 24
Population: ITT population (participants with concomitant statin therapy)
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W With Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W With Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin
Number analyzed (Participants) | 156 | 76 | 308
percent change | -0.1 (2.4) | -6.7 (3.3) | -15.2 (1.6)
Statistical Analysis 1: Comparison: Placebo Q2W With Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin; [analysis description as in outcome 33, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Robust — Threshold for significance ≤ 0.025; Adjusted Mean Difference = -15.1, 97.5% CI 2-sided [-21.5 to -8.6]

43. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides in Participants Not Receiving Concomitant Statin Therapy at Week 12 - ITT Analysis
Description: as for outcome 35
Time Frame: From Baseline to Week 12
Population: ITT population (participants without concomitant statin therapy)
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W Without Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W Without Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin
Number analyzed (Participants) | 71 | 37 | 144
percent change | 1.8 (3.2) | -18.3 (4.6) | -12.3 (2.3)
Statistical Analysis 1: Comparison: Placebo Q2W Without Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin; [analysis description as in outcome 33, analysis 1]; Test type: Superiority or Other; p = 0.0004, Regression, Robust — Threshold for significance ≤ 0.025; Adjusted Mean Difference = -14.1, 97.5% CI 2-sided [-22.9 to -5.2]

44. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides in Participants Receiving Concomitant Statin Therapy at Week 12 - ITT Analysis
Description: as for outcome 35
Time Frame: From Baseline to Week 12
Population: ITT population (participants with concomitant statin therapy)
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W With Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W With Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin
Number analyzed (Participants) | 156 | 76 | 308
percent change | 0.5 (2.4) | -7.3 (3.5) | -13.1 (1.7)
Statistical Analysis 1: Comparison: Placebo Q2W With Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin; [analysis description as in outcome 33, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Robust — Threshold for significance ≤ 0.025; Adjusted Mean Difference = -13.6, 97.5% CI 2-sided [-20.3 to -6.9]

45. Secondary Outcome: Percent Change From Baseline in Apo A1 in Participants Not Receiving Concomitant Statin Therapy at Week 24 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 24 from MMRM model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment. Subjects of the ITT population (subjects with or without concomitant statin therapy) with one baseline and at least one post-baseline Apo A1 value on- or off-treatment (Apo A1 ITT population). Alirocumab 75 mg Q2W arm (calibrator arm) was included only to facilitate comparison of results of this study with the results of other studies that used an alirocumab 75 mg Q2W regimen. Hence no statistical comparison was performed for this arm.
Time Frame: From Baseline to Week 24
Population: Apo A1 ITT population (participants without concomitant statin therapy)
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W Without Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W Without Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin
Number analyzed (Participants) | 71 | 34 | 138
percent change | -1.4 (1.3) | 3.1 (1.9) | 5.2 (0.9)
Statistical Analysis 1: Comparison: Placebo Q2W Without Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.025; LS Mean Difference = 6.6, 97.5% CI 2-sided [3.0 to 10.2]

46. Secondary Outcome: Percent Change From Baseline in Apo A1 in Participants Receiving Concomitant Statin Therapy at Week 24 - ITT Analysis
Description: as for outcome 45
Time Frame: From Baseline to Week 24
Population: Apo A1 ITT population (participants with concomitant statin therapy)
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W With Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W With Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin
Number analyzed (Participants) | 146 | 75 | 292
percent change | 2.9 (1.0) | 6.5 (1.4) | 5.5 (0.7)
Statistical Analysis 1: Comparison: Placebo Q2W With Concomitant Statin vs Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0306, Mixed Models Analysis — Threshold for significance ≤ 0.025; LS Mean Difference = 2.7, 97.5% CI 2-sided [-0.1 to 5.4] — Alirocumab 300 mg vs. Placebo

47. Secondary Outcome: Percent Change From Baseline in Apo A1 in Participants Not Receiving Concomitant Statin Therapy at Week 12 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment. Apo A1 ITT population (subjects with or without concomitant statin therapy). Alirocumab 75 mg Q2W arm (calibrator arm) was included only to facilitate comparison of results of this study with the results of other studies that used an alirocumab 75 mg Q2W regimen. Hence no statistical comparison was performed for this arm.
Time Frame: From Baseline to Week 12
Population: Apo A1 ITT population (participants without concomitant statin therapy)
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W Without Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W Without Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W Without Concomitant Statin
Number analyzed (Participants) | 71 | 34 | 138
percent change | -1.8 (1.3) | 2.4 (1.8) | 4.6 (0.9)

48. Secondary Outcome: Percent Change From Baseline in Apo A1 in Participants Receiving Concomitant Statin Therapy at Week 12 - ITT Analysis
Description: as for outcome 47
Time Frame: From Baseline to Week 12
Population: Apo A1 ITT population (participants with concomitant statin therapy)
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W With Concomitant Statin | Alirocumab 75 mg Q2W/Up 150 mg Q2W With Concomitant Statin | Alirocumab 300 mg Q4W/Up 150 mg Q2W With Concomitant Statin
Number analyzed (Participants) | 146 | 75 | 292
percent change | 2.7 (1.0) | 6.1 (1.4) | 6.0 (0.7)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (Week 56 post-treatment follow-up visit) regardless of seriousness or relationship to investigational product.
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during the 'treatment-emergent period' (the time from the first dose of study drug up to the last dose of study drug +70 days).
Groups:
- Placebo Q2W: Two SC injections of placebo (for alirocumab) Q2W with or without stable statin therapy for 48 weeks.
- Alirocumab 75 mg Q2W/Up 150 mg Q2W: One SC injection of Alirocumab 150 mg Q4W alternating with 2 SC injections of placebo Q4W with or without stable statin therapy for 48 weeks. Alirocumab dose up-titrated to 150 mg from Week 12 when LDL-C levels ≥ 70 mg/dL (1.81 mmol/L) (for very high CV risk subjects) or ≥ 100 mg/dL (2.59 mmol/L) (for moderate and high CV risk subjects) at Week 8.
- Alirocumab 300 mg Q4W/Up 150 mg Q2W: Two SC injections of Alirocumab 300 mg Q4W alternating with two SC injections of placebo Q4W with or without stable statin therapy for 48 weeks. Alirocumab dose up-titrated to 150 mg from Week 12 when LDL-C levels ≥ 70 mg/dL (1.81 mmol/L) (for very high CV risk subjects) or ≥ 100 mg/dL (2.59 mmol/L) (for moderate and high CV risk subjects) at Week 8.
Arm/Group | Placebo Q2W | Alirocumab 75 mg Q2W/Up 150 mg Q2W | Alirocumab 300 mg Q4W/Up 150 mg Q2W
Serious Adverse Events (participants affected / at risk) | 33/229 | 13/115 | 53/458
Other Adverse Events (participants affected / at risk) | 118/229 | 55/115 | 229/458
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Q2W (N=229) | Alirocumab 75 mg Q2W/Up 150 mg Q2W (N=115) | Alirocumab 300 mg Q4W/Up 150 mg Q2W (N=458)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 2
Angina pectoris (Cardiac disorders) | 1 | 1 | 1
Angina unstable (Cardiac disorders) | 2 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 2
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 2
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 3 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 | 0 | 0
Epiploic appendagitis (Gastrointestinal disorders) | 0 | 0 | 1
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal spasm (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1
Volvulus (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
Coronary artery restenosis (General disorders) | 1 | 0 | 0
Impaired healing (General disorders) | 0 | 0 | 1
Non-Cardiac chest pain (General disorders) | 1 | 1 | 4
Oedema peripheral (General disorders) | 0 | 1 | 0
Pelvic mass (General disorders) | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Acute hepatitis c (Infections and infestations) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 2 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Monarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Adrenocortical carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Intraductal papillary-mucinous carcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Cervical radiculopathy (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 2
Completed suicide (Psychiatric disorders) | 0 | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 1
Ureteric obstruction (Renal and urinary disorders) | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Prostatic obstruction (Reproductive system and breast disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0
Vascular compression (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Q2W (N=229) | Alirocumab 75 mg Q2W/Up 150 mg Q2W (N=115) | Alirocumab 300 mg Q4W/Up 150 mg Q2W (N=458)
Diarrhoea (Gastrointestinal disorders) | 17 | 4 | 25
Nausea (Gastrointestinal disorders) | 15 | 7 | 19
Injection site reaction (General disorders) | 16 | 10 | 74
Non-Cardiac chest pain (General disorders) | 5 | 6 | 7
Bronchitis (Infections and infestations) | 12 | 7 | 19
Nasopharyngitis (Infections and infestations) | 18 | 10 | 39
Sinusitis (Infections and infestations) | 11 | 4 | 28
Upper respiratory tract infection (Infections and infestations) | 18 | 8 | 41
Urinary tract infection (Infections and infestations) | 10 | 7 | 28
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 7 | 29
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 3 | 29
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13 | 4 | 10
Headache (Nervous system disorders) | 13 | 6 | 29
Hypertension (Vascular disorders) | 12 | 4 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Not less than 45 days prior to submission for publication or presentation, the Institution shall, or cause the Principal Investigator to, provide the Sponsor with a copy of the Manuscript. The Institution shall consider in good faith any comments from the Sponsor regarding the content, and shall delete Confidential Information upon written request of the Sponsor. At the Sponsor's request, the Institution shall delay publication for an additional 60 days to allow patent applications to be filed.